CLINICAL TRIAL: NCT04897087
Title: Openness and Learning Following Patient Safety Events: Involving Patients and Carers When Things go Wrong in Health Care a Qualitative Enquiry
Brief Title: Openness and Learning Joint Commission: Using Patient Experience for Improvement Following a Patient Safety Event
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NHS Education for Scotland (Other Government)
Responsible Party: Principal Investigator, Jean McQueen, Principal Educator, NHS Education for Scotland
Other Study IDs: 21/WS/0048
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Patient Safety
Keywords: openness and learning; adverse events; qualitative research
MeSH Terms: interventions — Risk Management

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: patient safety event — This study will explore the perceptions of patients, carers and relatives who have experienced a patient safety event. Telephone interviews will be undertaken lasting up to 60 minutes This study involves NHS patients, their carers or relatives. We will ask participants about their experience of being involved a patient safety event and the barriers and enablers to participation in the review. We will ask what 'good' patient involvement in patient safety reviews should look like from those with lived experience. This is because we wish to understand from their perspective what matters to them when things go wrong and how best to involve them.

SUMMARY:
The focus of our work is openness, learning and person-centred involvement following patient safety incidents in health care. We will explore patients, carers and relatives' perspectives on what is important to them, what facilitates and impedes their involvement in patient safety reviews and what matters to them. We are interested in exploring how patient, carer and relative involvement can assist reconciliation, organisational and national learning. Information gained will be used to support the development of national guidance around involving people in a compassionate and caring way and how their experience could help organisational and national learning when things go wrong in health care.

DETAILED DESCRIPTION:
INTRODUCTION:

Scotland is committed to a person-centred approach to social care and health services. This includes a duty of candour towards service users and families when things go wrong. Typical of service users and families who are involved in patient safety incidents or make complaints about services is the stated intent that they "don't want anyone else to go through what they have experienced". Inherent in this sentiment is the desire that services learn from feedback, safety incidents, complaints and near misses where unnecessary harm is caused (or could have been) when interacting with health care services. Current guidance suggests health and care providers offer an explanation of the incident, an apology, and a commitment to prevent recurrence. There is growing recognition among health care providers and policy makers that when things go wrong, the patient or their families should be heard and participate in the incident investigation process (Kok et al 2018). Guidance on how best to involve patients, carers and relatives in a caring and compassionate manner is lacking and current practice variable. The joint commission for openness and learning is committed to understanding and learning what 'good' patient involvement in patient safety reviews could look like as part of improving patient safety in health care.

AIMS:

This study is part of a larger programme of work being undertaken by NHS Education for Scotland (NES) and Health Improvement Scotland (HIS) on behalf of the Scottish Government. The focus of our work is openness, learning and person-centred involvement following patient safety incidents in health care. We will explore patients, carers and relatives' perspectives on what is important to them, what facilitates and impedes their involvement in patient safety reviews and what matters to them. We are interested in exploring how patient, carer and relative involvement can assist reconciliation, organisational and national learning. Information gained will be used to support the development of national guidance around involving people in a compassionate and caring way and how their experience could help organisational and national learning when things go wrong in health care.

OBJECTIVES:

* To identify factors that facilitate and impede patient, carer and relative involvement using patient perspectives to guide and strengthen how the NHS involves, communicates and learns with patients their carers and relatives
* To explore how to involve people in a compassionate and caring way and how their experience can be harnessed to assist national and organisational learning

ELIGIBILITY:
Inclusion Criteria:

* Patients or family members of patients who have experienced a serious health care incident/patient safety event in the last 10 years who reside in Scotland, are aged 18 years or over and speak English. We will exclude participants where an investigation or litigation claim is ongoing or have been involved in an incident that happened less than a year ago, where the investigation is still ongoing or who are currently involved in legal action related to the incident.

Exclusion Criteria:

* We will exclude participants where an investigation or litigation claim is ongoing or have been involved in an incident that happened less than a year ago, where the investigation is still ongoing or who are currently involved in legal action related to the incident.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients or family members of patients who have experienced a serious health care incident/patient safety event
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-05-20 (Estimated); Primary Completion 2022-01-20 (Estimated); Study Completion 2022-01-20 (Estimated)

PRIMARY OUTCOMES:
Qualitative data | 60 mins
  Telephone interviews lasting up to 60 minutes will be conducted by qualitative researchers

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Education for Scotland, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
National Report, Peer Review Journal publication
Supporting Information: Study Protocol
Time Frame: 05.01.22 for 6 weeks
URL: https://www.nes.scot.nhs.uk/our-work/person-centred-care/